CLINICAL TRIAL: NCT03052855
Title: Title: Inflammatory Biomarkers and Brain Metabolites, a Study Based on Magnetic Resonance Spectroscopy.
Brief Title: Inflammatory Biomarkers and Brain Metabolites, a Study Based on Magnetic Resonance Spectroscopy
Acronym: BICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF9741; 2016-A01267-44 (Other: Agence NAtionale de Sécurité du Médicament)
Record Dates: First submitted 2017-01-31; First posted 2017-02-14 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Depression
Keywords: Psychiatry; Suicidal behaviour; Cerebral metabolites; MRI; Inflammatory markers
MeSH Terms: conditions — Depression | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): All the participants of the 3 groups (depressed patients with suicide attempt, depressed patients without suicide attempt, healthy volunteers) will have to realize a MRI and biological samples.
  Interventions: Other: Magnetic Resonance Imaging (MRI) and biological samples

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) and biological samples — Participants will have to do a MRI and biological samples.

SUMMARY:
Suicidal behaviors (SB) are a major health problem in France : 10 000 suicides and 220 000 suicide attempts every year. SB management is therefore a major public health issue.

Evidence associated dysregulation of the serotonergic system and the hypothalamic-pituitary-adrenal axis to vulnerability to SB. Recent data point to linke these abnormalities with neuroinflammatory clues, glutamatergic function and neuronal plasticity. There is a need to better understand the physiopathology and develop diagnostic and therapeutic tools in SB.

The investigators hypothesize that increased peripheral biomarkers of inflammation would correlate to a disturbance of the cerebral metabolites, such as glutamate and NAA, especially in suicidal patients.

Our aim is to compare rates of cerebral metabolites, in particular the complex glutamine/glutamate, in cerebral areas involved in suicidal vulnerability (the anterior cingulate cortex and the orbito-frontal cortex) between person with unipolar disorder with and without suicidal attempt.

DETAILED DESCRIPTION:
69 patients : 23 with suicidal thoughts and attempt, 23 with suicidal thoughts without attempt and 23 healthy volunteers.

2 visits :

* Inclusion visit (V0) : (Day 1)

  o Clinical interview : self and hetero assessment questionnaire
* Visit V1 (as soon as possible, day 1 if available) :

  * MRI (spectroscopy)

ELIGIBILITY:
Non-specific inclusion criteria:

* Having signed informed consent
* Able to understand nature, aims and methodology of the study

Specific inclusion criteria :

* Suicidal patient with suicide attempt :

  * Persistent depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders - V (DSM-V) criteria, and evaluated by the Mini International Neuropsychiatric Interview (MINI)
  * Hamilton Depression Scale > 7
  * Suicide attempt < 1 week
* Suicidal patient without suicide attempt :

  * Persistent depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders - V (DSM-V) criteria, and evaluated by the Mini International Neuropsychiatric Interview (MINI)
  * Hamilton Depression Scale > 7
  * No history of suicide attempt
* Healthy volunteers :

  * No psychiatric history
  * No history of suicide attempt

Exclusion criteria:

* Actual somatic, neurological or inflammatory pathology (C-Reactive Protein > 10mg/L)
* Traumatic brain injury with loss of consciousness
* Antibiotic treatment or anti-inflammatory treatment
* Actual toxic abuse according to DSM-V (except tobacco and alcohol)
* Actual or passed history of psychotic disorder
* Patient on protective measures (guardianship or trusteeship)
* Deprived of liberty subject (judicial or administrative decision)
* Pregnant women or breastfeeding
* Contraindications to MRI scan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Glutamine (Glu) and Glutamate (Glx) levels | At V1 (the day of the MRI)
  Levels of Glu/Glx in the anterior cingulate cortex and the orbitofrontal cortex between the depressed patients with and without suicide attempt

SECONDARY OUTCOMES:
Link between rate of Interleukin 1, 2, 4, 5, 6, 7, 9, 10, 13 and suicide attempt | At V1 (the day of the MRI)
  Comparison of Interleukin 1, 2, 4, 5, 6, 7, 9, 10, 13 between the 3 groups
Level of N-Acetyl-Aspartate (NAA) | At V1 (the day of the MRI)
  Comparison of levels of NAA in the anterior cingulate cortex and the orbito-frontal cortex between the 3 groups
Level of Choline (Cho) | At V1 (the day of the MRI)
  Comparison of levels of Cho in the anterior cingulate cortex and the orbito-frontal cortex between the 3 groups
Level of Myo-inositol (Myo) | At V1 (the day of the MRI)
  Comparison of levels of Myo in the anterior cingulate cortex and the orbito-frontal cortex between the 3 groups
Level of Creatinine (Cr) | At V1 (the day of the MRI)
  Comparison of levels of Creatinine (Cr) in the anterior cingulate cortex and the orbito-frontal cortex between the 3 groups
Link between level of suicidal intentionality assessed by the Columbia Suicide Severity Rating Scale (CSS-RS) and metabolites levels | At V1 (the day of the MRI)
  Relationship between level of suicidal intentionality and Glu/Glx levels between the 3 groups
Link between level of depression assessed by the clinician with the Hamilton Rating Scale (HAMD) and metabolite levels | At V1 (the day of the MRI)
  Relationship between level of depression and Glu/Glx levels between the 3 groups
Link between level of depression self assessed with the Beck Scale and metabolites levels | At V1 (the day of the MRI)
  Relationship between level of depression and Glu/Glx levels between the 3 groups
Link between rate of Tumor necrosis factor alpha (TNF α) and suicide attempt | At V1 (the day of the MRI)
  Comparison of biomarkers inflammation (TNF α) between the 3 groups
Link between rate of Tumor necrosis factor beta (TNFβ) and suicide attempt | At V1 (the day of the MRI)
  Comparison of biomarkers inflammation (TNFβ) between the 3 groups
Link between rate of Interferon gamma (IFNγ) and suicide attempt | At V1 (the day of the MRI)
  Comparison of biomarkers inflammation (IFNγ) between the 3 groups
Link between rate of C-Reactive Protein (CRP) and suicide attempt | At V1 (the day of the MRI)
  Comparison of biomarkers inflammation (CRP) between the 3 groups
Link between rate of Interferon Gamma Inducing Factors (IGIF)and suicide attempt | At V1 (the day of the MRI)
  Comparison of biomarkers inflammation (IGIF) between the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric COPPOLA, MD, Principal Investigator — Montpellier Hospital University
Locations (1):
- Montpellier Hospital University, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olie E, Clain G, Malestroit M, Fiedos D, Cognasse F, Deverdun J, Bars EL, Courtet P. Association of Suicidal Status, Inflammation Markers, and Resting-State Functional Activity and Connectivity in Patients With Major Depressive Disorder. J Clin Psychiatry. 2024 Jun 26;85(3):23m15148. doi: 10.4088/JCP.23m15148. PMID 39874064